CLINICAL TRIAL: NCT00454623
Title: Normal Serum Adiponectin Levels in Females During the Childbearing Ages and Normal Serum Adiponectin Levels in Pregnancy
Brief Title: Normal Serum Adiponectin Levels in Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Cooper Health System (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06041EX
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2007-04-02 (Estimated); Status verified 2007-03

CONDITIONS: Diabetes Mellitus
Keywords: Adiponectin; diabetes; metabolism; Adiponectin levels
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: drawing serum adiponectin level

SUMMARY:
The purpose of the study is to establish the normal levels of the hormone adiponectin in women. Adiponectin is a newly discovered hormone, which is said to be associated with many changes in the human body and metabolism. The researchers aim is to establish the normal levels of this hormone. Hence, the researchers can identify people with abnormal levels who may be at risk of diseases and can do more studies to help them.

DETAILED DESCRIPTION:
The prevalence of obesity has increased dramatically in recent years . It is commonly associated with type 2 diabetes, coronary artery disease, and hypertension, and the coexistence of these diseases has been termed the metabolic syndrome. White Adipose Tissue (WAT) has been increasingly recognized as an important endocrine organ that secretes a number of biologically active "adipokines" . Of these adipokines, adiponectin has recently attracted much attention because of its antidiabetic and antiatherogenic effects and is expected to be a novel therapeutic tool for diabetes and the metabolic syndrome . Adiponectin directly regulates glucose metabolism and insulin sensitivity by activation of AMPK.

Adiponectin expression is reduced in obese, insulin-resistant rodent models. Plasma adiponectin levels are also decreased in an obese rhesus monkey model that frequently develops type 2 diabetes. Levels have also been reported to be reduced in obese humans, particularly those with visceral obesity, and to correlate inversely with insulin resistance. Prospective and longitudinal studies have shown that lower adiponectin levels are associated with a higher incidence of diabetes.

Hypoadiponectinemia has been demonstrated to be independently associated with the metabolic syndrome. Reduced plasma adiponectin levels are also commonly observed in a variety of states frequently associated with insulin resistance, such as cardiovascular disease, ischemic heart disease, and hypertension. In women, lower adiponectin levels were associated with breast cancer, endometrial cancer, and polycystic ovarian syndrome.

By establishing normal serum levels of Adiponectin, researchers will be able to demonstrate deviations from the norm associated with investigated diseases and variables. When applied to pregnancy, it will help identify obstetrical complications associated with abnormal levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 15 - 40 years old.
2. BMI: 18.5 - 24.9
3. No medical or chronic health problems.
4. If pregnant, singleton.
5. First blood sample can be obtained before 13 weeks gestation.
6. Plans to continue pregnancy till term and deliver at our hospital

Exclusion Criteria:

1. Hypertension.
2. Diabetes Mellitus.
3. Ischemic heart disease.
4. Metabolic disorders e.g. hyperlipidemia, hypercholesterolemia.
5. Endocrinological diseases e.g. thyroid or adrenal diseases.
6. Chronic Debilitating diseases e.g. SLE, or Cancer.
7. BMI less than18.5 or greater than 25.
8. Anorexia or Bulimia.
9. Polycystic ovarian disease.
10. In pregnant group:

    1. Multiple gestations.
    2. Hyperemesis or dehydration.
    3. History of Gestational Diabetes, Preeclampsia, or other complications with previous pregnancies
    4. If abnormal weight gain during pregnancy, will continue in the study but would not be included in establishing normal levels.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300
Dates: Start 2006-03; Study Completion 2007-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elshoreya, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

REFERENCES:
- [Background] Cseh K, Baranyi E, Melczer Z, Kaszas E, Palik E, Winkler G. Plasma adiponectin and pregnancy-induced insulin resistance. Diabetes Care. 2004 Jan;27(1):274-5. doi: 10.2337/diacare.27.1.274. No abstract available. PMID 14694004